CLINICAL TRIAL: NCT06365385
Title: Postprandial Metabolic and Appetite Responses to Different Food Intake Sequences in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Federação Portuguesa de Futebol (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FOODSEQ-MARS
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Nutrition, Healthy; Postprandial Hyperglycemia; Hunger; Craving
Keywords: food order; meal sequence; glucose metabolism; lipid metabolism; satiety; sport nutrition
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: This study is a randomised controlled trial with a counterbalanced crossover design. Block randomisation will be performed by an external researcher, and allocation concealment will be ensured through the use of sequentially numbered, opaque, sealed envelopes.
Who Masked: Outcomes Assessor
Masking Description: This is a non-blind trial, since both participants and the investigator delivering the test-meal will be able to see the ingredients and the order in which they are consumed. However, outcome assessors will be blinded to the intervention sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CL - CF (Experimental): The interventions (carbohydrate-last meal pattern (CL) or carbohydrate-first meal pattern (CF)) will be delivered in random order at two study visits, separated by a wash-out period of 7 days. If participants are allocated to this study arm, they will receive the CL on the first visit and the CF on the second visit.
  The nutritional composition of the test-meal will comply to the current sports nutrition guidelines for the pre-exercise meal (i.e., 1-4 g of CHO/kg of body mass, moderate amounts of protein, low-fat and fibre content, 5-10 mL/kg of body mass of fluids) (Thomas et al., 2016). Participants will be encouraged to consume the meal in full within 15 minutes, at a comfortable pace, to mimic real eating circumstances.
  Interventions: Other: Carbohydrate-last meal pattern; Other: Carbohydrate-first meal pattern
- CF - CL (Active Comparator): The interventions (carbohydrate-last meal pattern (CL) or carbohydrate-first meal pattern (CF)) will be delivered in random order at two study visits, separated by a wash-out period of 7 days. If participants are allocated to this study arm, they will receive the CF on the first visit and the CL on the second visit.
  The test-meal will be identical and isocaloric in both interventions of the study.
  Interventions: Other: Carbohydrate-last meal pattern; Other: Carbohydrate-first meal pattern

INTERVENTIONS:
Other: Carbohydrate-last meal pattern — Skyr yoghurt, whey protein and almonds over ~5 min, immediately followed by white bread, strawberry jam, banana and pulp-free orange juice over ~10 min.
  Other Names: CL; CHO-last
Other: Carbohydrate-first meal pattern — White bread, strawberry jam, banana and pulp-free orange juice over ~10 min, immediately followed by skyr yoghurt, whey protein and almonds over ~5 min.
  Other Names: CF; CHO-first

SUMMARY:
Emerging evidence suggests that following a 'carbohydrate-last meal pattern', wherein foods rich in protein, fat, fiber, and/or polyphenols are consumed before sources of simple carbohydrate (CHO) in a meal, results in reduced postprandial glycaemic responses than the reverse food order or a co-ingestion pattern. This effect has been observed across the spectrum of glucose tolerance, from patients with diabetes to individuals with normal glucose tolerance (Kuwata et al., 2016; Nishino et al., 2018; Lu et al., 2019; Sun et al., 2020). Furthermore, reduced glucose excursions have been linked to decreased subsequent hunger and energy intake (Lu et al., 2019; Wyatt et al., 2021).

However, to date, no studies on food intake sequence have targeted athletes, despite their increased CHO demands (Thomas et al., 2016) which could expose them to repeated episodes of hyperglycaemia and high glycaemic variability, known to increase the risk of adverse cardiovascular outcomes and all-cause mortality (Loader et al., 2015; Cavero-Redondo et al., 2017; Faerch et al., 2018). Additionally, athletes often face pressure to meet body composition standards and may benefit from strategies that enhance satiety and craving control. Finally, there is reason to believe that better glycaemic control could lead to improved performance, given that enhancements in endurance activities have been observed with a low-glycemic-index diet compared to a high-glycemic-index diet (Heung-Sang Wong et al., 2017).

Therefore, this randomised crossover trial is part of a wider project which seeks to explore the impact of food intake sequence on metabolic health and performance in athletes. Specifically, this trial aims to investigate the acute, postprandial metabolic and appetite responses to consuming an identical meal in two intake sequences (CHO-last versus CHO-first) in athletes, while in the resting state.

DETAILED DESCRIPTION:
Participants will be required to visit the research facilities at Cidade do Futebol (Portugal Football School's headquarters) on three separate occasions, following a 10-12-hour overnight fast and abstaining from alcohol consumption and strenuous physical activity the day before (e.g. no exercise causing sweating or heavy breathing). Visits will be separated by a wash-out period of 7 days to ensure participants experience similar dietary and physical activity patterns in the 24 hours preceding the trials. Each visit is expected to last approximately 4 hours.

In the screening and familiarisation visit, athletes will be asked to provide written informed consent to participate in the study and answer a series of questions to confirm their eligibility and safety for enrolment. Subsequently, an anthropometric assessment, blood pressure measurement, fasted blood collection and 2-hour 75-g oral glucose tolerance test (OGTT) will be performed to establish participants' baseline characteristics and analyse biochemical markers of the glucose and lipid metabolism to identify any further exclusion criteria (i.e., glycated haemoglobin (HbA1c); glucose; insulin; triglycerides; total, high-density lipoprotein and low-density lipoprotein cholesterol; haemogram and high-sensitivity C-reactive protein). To familiarise participants with the cannulation procedure ahead of the experimental trials, a trained and experienced nurse will insert a cannula (a small plastic tube) into a vein on the participants' arm, from which fasting and 2-h OGTT blood samples will be drawn (15 ml in total).

Eligible participants will be instructed to monitor their diet and physical activity for 24 hours before their first experimental visit and replicate these patterns before the second experimental visit.

In both experimental visits, participants will arrive at the research facilities between 8:00-9:00 and rest comfortably for 10 minutes. Body mass and blood pressure will be remeasured. Then, cannulation will be performed, and 18.5 ml venous blood samples will be drawn immediately before and at 30, 60, 90, 120, and 180 minutes after the meal challenge to assess postprandial changes in insulin, glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP), ghrelin, peptide YY (PYY), triglycerides, and non-esterified fatty acids (NEFA) concentrations. At similar timepoints, as well as at 15 and 45 minutes, capillary blood glucose will be measured using a finger prick glucometer, and appetite ratings will be marked by the athletes on 100-mm visual analogue scales.

Upon completing the research assessments, participants will be asked to photograph and record the timing, type, and amounts of foods, drinks, and/or supplements consumed for an additional 3 hours to evaluate their prospective, ad libitum intake.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-64 years old)
* Male
* Trained (meeting training and performance caliber criteria ≥Tier 2; McKay et al., 2022)
* Healthy (meeting the exclusion criteria for medical conditions)
* Normal glucose tolerant according to the latest criteria established by the American Diabetes Association (ElSayed et al., 2023): HbA1c <5.7%, fasting plasma glucose <5.6 mmol/L (100 mg/dL) and 2-h plasma glucose <7.8 mmol/L (140 mg/dL) during a 75-g OGTT
* Able and willing to provide informed consent and safely comply with study procedures

Exclusion Criteria:

* Any medical condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias into the experiment (e.g. anaemia and other haematological disorders; alcohol or substance abuse; any condition affecting the glucose and lipid metabolism or appetite, reviewed on a case by case basis)
* Any reported medication or supplementation that may interfere with the glucose metabolism (e.g., acarbose, insulin, metformin, semaglutide, thiazolidinediones, sulfonylureas, corticosteroids, thiazide diuretics); lipid metabolism (e.g., statins, nicotinic acid, colestyramine anhydrous, ezetimibe, fibrates, L-carnitine); or appetite (e.g., metoclopramide, carbamazepine, phenobarbital, phenytoin, primidone). Other medication and supplementation will be reviewed on a case by case basis.
* Known food allergy, intolerance or hypersensitivity to any of the test-meal ingredients
* Recent change in body mass (± 2 kg in the last 2 months)
* Smoking
* Having donated more than 400 ml of blood within 3 months of the screening visit or more than 1500ml of blood in the previous 12 months

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose concentrations | Baseline and 15, 30, 45, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the incremental area under the curve 0-120 and 0-180 min; peak concentrations (mmol/L); time-to-peak (min); and change from baseline data (mmol/L) of capillary blood glucose measured by a validated glucometer

SECONDARY OUTCOMES:
Postprandial subjective appetite ratings | Baseline and 15, 30, 45, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the total area under the curve 0-180 min; peak/nadir rating (mm); time-to-peak/nadir (min); and change from baseline data (mm) of appetite ratings measured by validated 100-mm visual analogue scales (Flint et al, 2000)
Prospective ad libitum energy intake | 0-3 hours post-trial
  Difference between food intake sequences in the total energy (kcal) consumed within 3 hours from the end of the experimental visit, assessed by a photography-supported dietary record of foods and fluids
Prospective ad libitum nutritional intake | 0-3 hours post-trial
  Difference between food intake sequences in the total carbohydrate, protein and fat (grams; g/kg of body mass and % of total energy intake) consumed within 3 hours from the end of the experimental visit, assessed by a photography-supported dietary record of foods and fluids
Postprandial serum insulin concentrations | Baseline and 30, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the incremental area under the curve 0-120 and 0-180 min; peak concentrations (microIU/ml); time-to-peak (min); and change from baseline data (microIU/ml) of serum insulin measured by a chemiluminescent immunoassay
Postprandial plasma total GLP-1 concentrations | Baseline and 30, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the incremental area under the curve 0-120 and 0-180 min; peak concentrations (pg/ml); time-to-peak (min); and change from baseline data (pg/ml) of plasma GLP-1 measured by a total GLP-1 ELISA kit
Postprandial plasma total GIP concentrations | Baseline and 30, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the incremental area under the curve 0-120 and 0-180 min; peak concentrations (pg/ml); time-to-peak (min); and change from baseline data (pg/ml) of plasma GIP measured by a total GIP ELISA kit
Postprandial serum total ghrelin concentrations | Baseline and 30, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the total area under the curve 0-120 and 0-180 min; nadir concentrations (pg/ml); time-to-nadir (min); and change from baseline data (pg/ml) of serum ghrelin measured by a total ghrelin ELISA kit
Postprandial plasma total PYY concentrations | Baseline and 30, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the incremental area under the curve 0-120 and 0-180 min; peak concentrations (pg/ml); time-to-peak (min); and change from baseline data (pg/ml) of plasma PYY measured by a total PYY ELISA kit
Postprandial serum triglyceride concentrations | Baseline and 30, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the incremental area under the curve 0-180 min; peak concentrations (mmol/L); time-to-peak (min); and change from baseline data (mmol/L) of serum triglycerides measured by the GPO/POD method
Postprandial serum NEFA concentrations | Baseline and 30, 60, 90, 120, 180 minutes following the test meal
  Difference between food intake sequences in the total area under the curve 0-180 min; nadir concentrations (mmol/L); time-to-nadir (min); and change from baseline data (mmol/L) of serum NEFA measured by an enzymatic colorimetric assay

CONTACTS AND LOCATIONS:
Overall Officials: Rita Giro, Principal Investigator — FCNAUP, University of Porto; Portugal Football School, Federação Portuguesa de Futebol
Locations (1):
- Cidade do Futebol, Avenida das Seleções, Oeiras, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No